CLINICAL TRIAL: NCT05018572
Title: Personalised Internet-based Treatment From a Biopsychosocial Perspective for Migraine Patients and Its Feasibility in Primary Care
Brief Title: Digital Treatment for Migraines - a Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VGFOUSA-963615
Record Dates: First submitted 2021-07-28; First posted 2021-08-24 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2022-10

CONDITIONS: Migraine With Aura; Migraine Without Aura
MeSH Terms: conditions — Migraine with Aura; Migraine without Aura

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The groups are predetermined based on the tool randomizer.org and blinded to the researcher assigning the participants to groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalised internet-based treatment "I am" (Experimental): Personalised internet-based treatment "I am".
  Interventions: Behavioral: I AM
- Treatment As Usual (No Intervention): Treatment in primary care / Treatment As Usual (TAU), which is medical treatment

INTERVENTIONS:
Behavioral: I AM — "I am" has a biopsychosocial perspective with a focus on pain management in migraines. The cognitive behavioural interventions being tested are Mindfulness, Acceptance and Commitment Therapy (ACT), Compassion Focused Therapy and Physiotherapist-led cardiotherapy. The treatment program consists of ten modules of texts, animated films with a fictional person to identify with, recorded audio exercises adapted for patients with migraines and filmed physiotherapeutic exercises with physiotherapists.The interventions in "I am" are personalised in that the first three modules and module 10 are for those who are being helped by a shorter treatment. The other modules, four to ten, are a more in-depth treatment for those who have frequent or chronic migraines. The participants are in contact with processors via message function as well as via phone at startup, at the middle of treatment and termination. The duration of treatment is 4-10 weeks.
  Other Names: Learn to live with migraines
  Arms: Personalised internet-based treatment "I am"

SUMMARY:
An individualised internet-based treatment from a biopsychosocial perspective for patients with migraines in primary care has been developed within the Vastra Gotaland region in 2019. The treatment program is called Learning to live with migraines, and goes by the acronym "I am" (Internet Approach to Migraine). In a pilot study, the treatment programme and its feasibility in primary care will be evaluated. It is hoped that the intervention "I am" can educate patients about their illness and help the patient manage migraine attacks so that the likelihood of difficulty and frequency of migraine attacks does not increase, as well as provide an increased function and quality of life.

DETAILED DESCRIPTION:
Purpose The overall purpose of the study is to evaluate in a pilot study the practical feasibility of a future randomized study to evaluate personalized digital biopsychosocial treatment method, "I am"- Learning to live with migraines in primary care.

Issues

Will a large or small percentage of individuals who are asked to participate in the study accept participation? Will the random advantage to the different groups make potential participants hesitant? Will measuring the effect be practicable? What investigative instruments are appropriate in this situation? Is a new investigative instrument to be built? Are the interventions reasonable to apply given the resources we can expect to have in a larger study? Will a large or small proportion of patients discontinue participation in the study for various reasons? How common are unforeseen problems (which may justify the exclusion of a patient or the negative/harmful effects of the intervention)? What change in endpoints is seen in the different groups?

ELIGIBILITY:
Inclusion Criteria:

* Women and men
* Age18 to 65
* Diagnosis migraine with (G43.0) or without aura (G43.1)
* 3-15 migraine days a month
* Access to computer/tablet or smartphone with bankid and internet connection

Exclusion Criteria:

* Ongoing malignant disease
* Other migraine diseases
* Moderate to severe psychiatric problems such as depression or anxiety disorder
* Neuropsychiatric conditions
* Psychosis disorders
* Addiction
* Personality disorders
* People who cannot read, speak or understand the Swedish language
* Ongoing psychological/psychotherapeutic treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2022-10-14 (Actual)

PRIMARY OUTCOMES:
Migraine Diary - change through week 2-10, and to 3 months follow up | Week 2-10 through the study and by 3 months follow up. The participant fills in a new form of the diary for each new attack.
  Frequency and severity of migraine attacks monthly: will take place via a Migraine Diary. Questions to answer; Migraine pain signal?
  When, day and time?
  Where does it hurt? Tick: Right temple, Left temple, Neck Inside the head, Area around the eye , other
  How's the pain? (Pulsating, burning, stinging, idling, stabbing)
  Strength, pain? (0-10)
  discomfort? (0-10)
  How do I try to deal with the pain? What emergency medication did you take at the beginning of the migraine attack?
  How long did the migraine attack last?
  Pain peak (throughout migraine attack) 0-10
  In total, how much emergency medicine have you taken throughout the migraine attack?
  Pre symptoms or other symptoms?
Employment rate - change through week 1, week 10, and by 3 months follow up | Week 1, week 10 and by 3 months follow up
  Employment rate: measured in percent by questions put to the participant.
Bulls eye - activation in valued direction -change through week 1 and week 10, and to 3 months follow up | Week 1-10 through the study and by 3 months follow up
  Measured with a Swedish version of Bulls eye (Lundgren, Louma, Dahl, Strohsal & Melin, 2012). ) The self-assessment scale is divided into four value areas in people's lives: work/education, leisure, relationships and self-care/health. The instrument has demonstrated a test-retest reliability of 0.86 and good criterion validity (Lundgren, Dahl & Hayes, 2008)

SECONDARY OUTCOMES:
Mental Health Continuum Short Form - Mental health and quality of life | Week 1 and week 10 and by 3 months follow up
  Measured with Mental Health Continuum Short Form (MHC-SF). The self-assessment form consists of 14 questions that focus on emotional, psychological and social well-being and are considered to have good psychometric properties (Keyes, 2005).
CORE-10 - A broader measure of mental health in terms of well-being, symptoms, function and risks | Week 1 and week 10 and by 3 months follow up
  Measured with the Swedish version CORE-10. The self-assessment form consists of 10 questions, one of which measures suicidality (Elfström, M. L., Evans, C., Lundgren, J., Johansson, B., Hakeberg, M., & Carlsson, S. G. (2012).
  Validation of the Swedish version of the Clinical Outcomes in Routine Evaluation Outcome Measure (CORE). Clinical Psychology and Psychotherapy. Epub ahead of print. doi:10.1002/cpp.1788)
Self-Efficacy for Exercise Scale - in their ability to conduct physical exercise | Week 1, week 5, week 10 and by 3 months follow up
  Measured by the Swedish version of the Self-Efficacy for Exercise Scale (SEE-EN). The form contains nine questions about the patient's faith in broad physical activity under different circumstances. A sum is calculated between 0 and 90, where higher number means higher confidence.Resnick B, Jenkins L 2000 Testing the reliability and validity of the Self-efficacy for Exercise Scale. Nursing Research 49: 149-159).The form has been translated into Swedish and tested for validity and reliability for patients with heart disease (Cavrak A 2010 Test of the psychometric properties of the Swedish version of the Self-Efficacy for Exercise scale for patients in cardiac rehabilitation.
  Masters Thesis, Uni-versity of Gothenberg.) And patients with long-term pain (Dahlbäck A, Andréll P, Varkey E. Reliability and Validity of the Swedish Version of the Self-Efficacy for Exercise Scale (SEE-SV) for Patients with Chronic Pain .2020 Unpublished manuscript).
Five Facet Mindfulness Questionnaire - conscious | Week 1, week 5, week 10 and by 3 months follow up
  Measured using the Swedish version of the Five Facet Mindfulness Questionnaire (FFMQ_SWE). FFMQ originally created by Baer et al. (2006) is a self-assessment form that aims to measure the ability to conscious presence. FFMQ_SWE consists of 29 claims and can be estimated between 1-5 points. The higher the score, the higher the self-rated ability to conscious presence. The internal validity and reliability of FFMQ_SWE is good (Lilja et al., 2011).
Self-Compassion Scale - Self compassion | Week 1, week 5, week 10 and by 3 months follow up
  Measured with Self-Compassion Scale - Short Form (SCS-SF). SCS-SF consists of 12 statements and is an abbreviated version of Self compassion scale (Neff, KD (2003b). The development and validation of a scale to measure self-compassion. Self & Identity, 2 (3), 223-250. doi: 10.1080 / 15298860309027. Self-compassion is measured with a corpse scale between 1 (almost never) and 5 (almost always) and has 6 subscales. SCS-SF has been shown to have good internal consistency (α ≥ .86) and constructivevalidity as it correlates positively with SCS (r ≥ 0.97). However, the subscale score has been shown to have poorer internal consistency and SCS-SF is therefore only suitable for measuring general self-compassion (Raes et al., 2011). Swedish translation of SCS-SF has been shown to have moderate internal consistency (α ≥ .68) (Almqvist & Johansson, 2016).
Exercise diary, condition | Week 1-10 through the study and by 3 months follow up
  Cardio training is measured with exercise diary Exercise diary contains filling in; activity, date, set
Two questions to Haskell 2007 - Physical activity | Week 1-10 through the study and by 3 months follow up
  Physical activity issues according to Haskell 2007. Two questions. Five total points or more means that the physical activity level is considered regular and corresponds to the public health recommendation. Below 5 total points means that the physical activity level needs to be increased.
Acceptance of the treatment | Week 10 and by 3 months follow up
  Measured with its own constructed form developed for the study. The form consists of four questions: Would you recommend the processing to someone else? How meaningful have you experienced the treatment scale 1-7, as well as two open questions answered in writing: what have you got out of the treatment? What has been less good about the treatment?

CONTACTS AND LOCATIONS:
Locations (1):
- FoU primary care Södra Älvsborg, Borås, Sven Eriksonsplatsen 4, Sweden